CLINICAL TRIAL: NCT04383678
Title: Outcome of COVID-19 Patients After Extracorporeal Membrane Oxygenation for Acute Respiratory Distress Syndrome: A Multicenter European Study
Brief Title: Outcome of COVID-19 Patients After Extracorporeal Membrane Oxygenation for Acute Respiratory Distress Syndrome
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Fausto Biancari, Professor, Helsinki University Central Hospital
Other Study IDs: COVID-19 ECMO
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: COVID-19; Extracorporeal Membrane Oxygenation Complication; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome | interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 positive patients
  Interventions: Device: Extracorporeal membrane oxygenation

INTERVENTIONS:
Device: Extracorporeal membrane oxygenation — Veno-venous or veno-arterial extracorporeal oxygenation

SUMMARY:
This study aims to investigate outcomes and predictors of outcome after extracorporeal membrane oxygenation (ECMO) therapy for severe acute respiratory syndrome (ARDS) in COVID-19 patients.

DETAILED DESCRIPTION:
We evaluated the outcome of adult patients with coronavirus disease 2019 (COVID-19)-related acute respiratory distress syndrome (ARDS) requiring the use of extracorporeal membrane oxygenation (ECMO).

ELIGIBILITY:
Inclusion Criteria:

* PCR-confirmed or suspected COVID-19 infection with ARDS who require any ECMO therapy

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with PCR-confirmed or suspected COVID-19 infection with ARDS who require veno-venous or veno-arterial ECMO therapy
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | Immediately after the intervention/procedure/surgery
  All-cause mortality

SECONDARY OUTCOMES:
Death on ECMO | During the intervention/procedure/surgery
  Death during ECMO therapy
Stroke | Immediately after the intervention/procedure/surgery
  Stroke was defined as any focal or global neurological syndrome caused by ischemia and/or hemorrhage not resolving within 24 hours.
Blood stream infection | Immediately after the intervention/procedure/surgery
  Blood stream infection detected on blood cultures
Lung complications requiring surgical treatment | Immediately after the intervention/procedure/surgery
  Pneuthorax, pneumonia and/or abscess requiring surgical treatment
Blood transfusion | Immediately after the intervention/procedure/surgery
  Transfusion of red blood cells
Acute kidney injury | Immediately after the intervention/procedure/surgery
  Acute renal failure according to the Kidney Disease: Improving Global Outcomes classification (KDIGO) criteria
Duration of mechanical ventilation | During index hospital stay follow-up until 1 year after ECMO initiation
  Duration of mechanical ventilation
Deep vein thrombosis | Immediately after the intervention/procedure/surgery
  Thrombosis of lower limb deep venous system
Pulmonary embolism | Immediately after the intervention/procedure/surgery
  Pulmonary embolism
Length of intensive care unit stay | Immediately after the intervention/procedure/surgery
  Length of stay in the intensive care unit
Length of hospital stay | Immediately after the intervention/procedure/surgery
  Length of hospital stay
Death after hospital discharge | Up to 6 months
  All-cause death

CONTACTS AND LOCATIONS:
Overall Officials: Fausto Biancari, Professor, Principal Investigator — Helsinki University Central Hospital
Locations (11):
- Helsinki University Hospital, Helsinki, Finland
- France (4):
  - University Hospital Jean Minjoz, Besançon
  - Nancy University Hospital, Nancy
  - Henri Mondon Unoversity Hospital, Paris
  - Robert Debré University Hospital, Reims
- Germany (2):
  - Hamburg University Heart Center, Hamburg
  - Münster University Hospital, Münster
- Italy (2):
  - S. Orsola Hospital, Bologna
  - Lecco Hospital, Lecco
- Karolinska University Hospital, Stockholm, Sweden
- University Hospitals of Leicester, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Biancari F, Mariscalco G, Dalen M, Settembre N, Welp H, Perrotti A, Wiebe K, Leo E, Loforte A, Chocron S, Pacini D, Juvonen T, Broman LM, Perna DD, Yusuff H, Harvey C, Mongardon N, Maureira JP, Levy B, Falk L, Ruggieri VG, Zipfel S, Folliguet T, Fiore A. Six-Month Survival After Extracorporeal Membrane Oxygenation for Severe COVID-19. J Cardiothorac Vasc Anesth. 2021 Jul;35(7):1999-2006. doi: 10.1053/j.jvca.2021.01.027. Epub 2021 Jan 19. PMID 33573928